CLINICAL TRIAL: NCT05475873
Title: Ondansetron for Postspinal Anesthesia Hypotension in Patients Undergoing Cesarean Section: A Randomized, Controlled Trial
Brief Title: Ondansetron for Postspinal Anesthesia Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2022-1
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-06

CONDITIONS: Adverse Effect
Keywords: Ondansetron; Coload; Hypotension; Cesarean section
MeSH Terms: conditions — Hypotension | interventions — Saline Solution; Ondansetron; Serotonin 5-HT3 Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Sham Comparator): A bolus of normal saline (2 ml) by IV was given 5 min before spinal anesthesia.
  Interventions: Drug: normal saline
- Ondansetron 4 mg (Experimental): A bolus of ondansetron (2 ml; 4mg) by IV was given 5 min before spinal anesthesia.
  Interventions: Drug: Ondansetron 4 mg
- Ondansetron 8 mg (Experimental): A bolus of ondansetron (2 ml; 8mg) by IV was given 5 min before spinal anesthesia.
  Interventions: Drug: Ondansetron 8 mg

INTERVENTIONS:
Drug: normal saline — A bolus of normal saline (2 ml) by IV was given 5 min before spinal anesthesia.
  Other Names: NS
  Arms: Control group
Drug: Ondansetron 4 mg — A bolus of ondansetron (2 ml; 4mg) by IV was given 5 min before spinal anesthesia.
  Other Names: 5-HT3 receptor antagonist
  Arms: Ondansetron 4 mg
Drug: Ondansetron 8 mg — A bolus of ondansetron (2 ml; 8mg) by IV was given 5 min before spinal anesthesia.
  Other Names: 5-HT3 receptor antagonist
  Arms: Ondansetron 8 mg

SUMMARY:
The purpose of this study is to investigate the effectiveness of ondansetron for postspinal anesthesia hypotension in patients undergoing cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Ondansetron have been highly demonstrated for prevention and/or treatment of post-spinal anesthesia hypotension. However, whether ondansetron could further reduction the incidence of post-spinal anesthesia hypotension is still unknown. The purpose of this study is to investigate the effectiveness of ondansetron for postspinal anesthesia hypotension in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Primipara or multipara
* Singleton pregnancy ≥ 37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥ 160mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-06-18 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Overall stability of systolic blood pressure control versus baseline | 1-15 minutes after spinal anesthesia
  Evaluated by performance error (PE)
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline

SECONDARY OUTCOMES:
Overall stability of heart rate control versus baseline | 1-15 minutes after spinal anesthesia
  Evaluated by performance error (PE).
The incidence of severe post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia
  Heart rate < 55 beats/min.
The incidence of hypertension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen | Immediately after delivery
  From umbilical arterial blood gases.
Base excess | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin R, Xu X, Zhao N, Shi Y, Chen Y, Chen J, Ni X. Effect of different prophylactical doses of ondansetron for the hemodynamic stability in patients undergoing cesarean section: a randomized controlled study. Front Med (Lausanne). 2025 Apr 3;12:1495721. doi: 10.3389/fmed.2025.1495721. eCollection 2025. PMID 40248081